CLINICAL TRIAL: NCT00770861
Title: A Multicenter, Prospective, Randomized, Double-blind, Placebo-Controlled, Dose-Titration Study of Nebivolol Monotherapy in Hispanic Patients With Stage 1 or Stage 2 Hypertension
Brief Title: A Study on the Efficacy and Safety of Nebivolol Monotherapy in Hispanic Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: John Whalen, MD, Executive Director, Clinical Development, Cardiovascular, Forest Research Institute, a Subsidiary of Forest Laboratories Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB-MD-16
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2011-01-26 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2010-12

CONDITIONS: Hypertension
Keywords: nebivolol; Bystolic ™; Hypertension; Hispanic; Hypertension in Hispanic patients
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol (Active Comparator): Nebivolol 5 mg, 5-mg Nebivolol nontrade tablets, oral administration ; Nebivolol 10 mg, 10-mg Nebivolol nontrade tablets, oral administration ; Nebivolol 20 mg, 20-mg Nebivolol nontrade tablets, oral administration ; Nebivolol 40 mg, two 20-mg Nebivolol nontrade tablets, oral administration
  Interventions: Drug: Nebivolol
- Placebo (Placebo Comparator): Matching placebo tablets, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nebivolol — Nebivolol 5 mg, 5-mg Nebivolol nontrade tablets , oral administration Nebivolol 10 mg, 10-mg Nebivolol nontrade tablets , oral administration Nebivolol 20 mg, 20-mg Nebivolol nontrade tablets , oral administration Nebivolol 40 mg, two 20-mg Nebivolol nontrade tablets , oral administration
  Other Names: Bystolic (TM)
  Arms: Nebivolol
Drug: Placebo — Matching placebo tablets, oral administration
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of nebivolol monotherapy in Hispanic patients with stage 1 or stage 2 hypertension

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18 to 80 years of age, self-identified as Hispanic or Latino ethnicity
* Females must be post-menopausal, or not pregnant and using an approved contraceptive regimen
* Meet criteria for stage I or II hypertension
* Currently not treated, or being treated with no more than two anti-hypertensive medications

Exclusion Criteria:

* Secondary hypertension
* Are taking three or more antihypertensive agents
* Have uncontrolled or poorly controlled diabetes mellitus type I or type II
* Evidence of other concurrent disease or conditions that might interfere with the conduct of the study
* Participation in any investigational study within 30 days of Screening (Visit 1).
* Have a history of hypersensitivity to nebivolol or other β-blockers, or any contraindication to β-blocker use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2008-09; Primary Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Lukic, MD., M.Sc., Study Director — Forest Research Institute, a subsidiary of Forest Laboratories Inc.
Locations (26):
- United States (23):
  - Forest Investigative Site, Buena Park, California
  - Forest Investigative Site, Chino, California
  - Forest Investigative Site, Long Beach, California
  - Forest Investigative Site, Los Angeles, California
  - Forest Investigative Site, National City, California
  - Forest Investigative Site, San Bernardino, California
  - Forest Investigative Site, Temecula, California
  - Forest Investigative Site, Tustin, California
  - Forest Investigative Site, Coral Gables, Florida
  - Forest Investigative Site FL2, Hialeah, Florida
  - Forest Investigative Site, Hialeah, Florida
  - Forest Investigative Site, Kissimmee, Florida
  - Forest Investigative Site, Miami, Florida
  - Forest Investigative Site, Pembroke Pines, Florida
  - Forest Investigative Site, West Palm Beach, Florida
  - Forest Investigative Site, Atlanta, Georgia
  - Forest Investigative Site, New Windsor, New York
  - Forest Investigative Site, The Bronx, New York
  - Forest Investigative Site, Carrollton, Texas
  - Forest Investigative Site, Corpus Christi, Texas
  - Forest Investigative Site, Dallas, Texas
  - Forest Investigative Site, El Paso, Texas
  - Forest Investigative Site, San Antonio, Texas
- Puerto Rico (3):
  - Forest Investigative Site, Ponce
  - Forest Investigative Site, Salinas
  - Forest Investigative Site, Santurce

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was one year, from November 2008 to November 2009, occurring at 29 centers in the US and 3 centers in Puerto Rico.
Pre-assignment Details: All patients went through a 4 week, single blind, placebo run-in/washout phase before randomization.
Period: Overall Study
Arm/Group | Nebivolol | Placebo
Started | 141 | 136
Completed | 131 | 120
Not Completed | 10 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Placebo | Total
Number analyzed (Participants) | 141 | 136 | 277
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 135 | 129 | 264
  >=65 years | 6 | 7 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 50.4 (8.7) | 50.4 (8.7) | 50.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 51 | 113
  Male | 79 | 85 | 164
Region of Enrollment [Number; unit: participants]
  United States | 134 | 131 | 265
  Puerto Rico | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Seated DBP at Week 8(LOCF).
Description: The primary efficacy parameter was the change from baseline in mean trough seated DBP at Week 8. The average of three consecutive BP measurements would be the mean trough seated DBP value.
Time Frame: From baseline visit 7 (week 0) to end of double-blind treatment phase visit 11 (week 8)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 141 | 135
mm Hg | -11.1 (8.8) | -7.3 (8.9)
Statistical Analysis 1: Comparison: Nebivolol vs Placebo; H0 - There was no difference in BP reduction between Neb and Placebo. The efficacy analyses were based on the ITT population for the double-blind treatment phase. The LOCF was used to impute missing postbaseline values. Sensitivity analyses were based on observed cases for all efficacy parameters. All statistical tests were two-sided hypothesis tests performed at the 5% level of significance for main effects. All confidence intervals were two-sided 95% confidence intervals; Test type: Superiority or Other; p < 0.0001, ANCOVA; Between-treatment comparison of efficacy was performed by ANCOVA, with treatment, baseline BMI, center as factors & baseline value as a covariate

2. Secondary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure (SBP) at Week 8 (LOCF).
Description: The secondary efficacy parameter was the change from baseline in mean trough seated SBP at Week 8. The average of three consecutive BP measurements would be the mean trough seated SBP value.
Time Frame: From baseline visit 7 (week 0) to end of double-blind treatment phase visit 11 (week 8)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 141 | 135
mm Hg | -14.1 (12.7) | -9.3 (13.0)
Statistical Analysis 1: Comparison: Nebivolol vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for a period of thirteen months, from November 2008 to December 2009.
Arm/Group | Nebivolol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/141 | 1/136
Other Adverse Events (participants affected / at risk) | 5/141 | 8/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=141) | Placebo (N=136)
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=141) | Placebo (N=136)
Headache (Nervous system disorders) | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & can embargo communications re: results for 60 days from time submitted to sponsor for review. PI shall not disclose sponsor's confidential information. Upon sponsor's request, PI shall delete any proprietary info & shall not include raw data in the publication. On sponsor's request, PI shall delay submission for any pub while sponsor files patent applications. Any publication will give recognition to Sponsor's support.